CLINICAL TRIAL: NCT01472237
Title: Randomized Cotrolled Trial of Nutritional Intervention Program in Malnourished (Mini Nutritional Assessment < 17) Patients Admitted for Heart Failure
Brief Title: Nutritional Intervention Program in Malnourished Patients Admitted for Heart Failure
Acronym: PICNIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Randomization was stopped early because a significant beneficial effect of nutritional intervention was found in the interim analysis
Sponsor: Hospital San Juan de la Cruz (Other)
Responsible Party: Principal Investigator, Juan Luis Bonilla Palomas, Cardiologist, Hospital San Juan de la Cruz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PICNIC-2011
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure; Malnutrition; Nutritional Intervention; Mortality
MeSH Terms: conditions — Heart Failure; Malnutrition

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Nutritional intervention (Active Comparator): It will last 6 months. Will be conducted by a physician nutrition specialist assisted by a technician in diet and nutrition. The first visit will take place during admission. The patient receives dietary advice and a customized diet designed to optimize energy intake and macro/micro-nutrients needs.
  Interventions: Other: Nutritional intervention
- Care as usual (Placebo Comparator): The patients are referred to their cardiologyst and primary care physicians
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — Modification of diet

SUMMARY:
The purpose of this study is to determine whether a modification of the diet of malnourished patients admitted for heart failure is beneficial in term of mortality,hospitalizations and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for heart failure
* > 18 years old
* Malnutrition determined by MNA test (< 17 points)

Exclusion Criteria:

* If is not possible to perform a nutritional assessment
* Planned PCI or CABG to correct heart failure etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Mortality and heart failure hospitalizations | 12 months

SECONDARY OUTCOMES:
Quality of life | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Juan de la Cruz, Úbeda, Jaen, Spain

REFERENCES:
- [Background] Bonilla-Palomas JL, Gamez-Lopez AL, Anguita-Sanchez MP, Castillo-Dominguez JC, Garcia-Fuertes D, Crespin-Crespin M, Lopez-Granados A, Suarez de Lezo J. [Impact of malnutrition on long-term mortality in hospitalized patients with heart failure]. Rev Esp Cardiol. 2011 Sep;64(9):752-8. doi: 10.1016/j.recesp.2011.03.009. Epub 2011 Jun 8. Spanish. PMID 21652135
- [Derived] Baldwin C, de van der Schueren MA, Kruizenga HM, Weekes CE. Dietary advice with or without oral nutritional supplements for disease-related malnutrition in adults. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002008. doi: 10.1002/14651858.CD002008.pub5. PMID 34931696
- [Derived] Bonilla-Palomas JL, Gamez-Lopez AL, Castillo-Dominguez JC, Moreno-Conde M, Lopez Ibanez MC, Alhambra Exposito R, Ramiro Ortega E, Anguita-Sanchez MP, Villar-Raez A. Nutritional Intervention in Malnourished Hospitalized Patients with Heart Failure. Arch Med Res. 2016 Oct;47(7):535-540. doi: 10.1016/j.arcmed.2016.11.005. PMID 28262195